CLINICAL TRIAL: NCT06899113
Title: Correlating Multispectral Near-Infrared Imaging to Standard Vascular Diagnostics
Status: Recruiting | Type: Observational
Sponsor: MIMOSA Diagnostics Inc. (Industry)
Collaborators: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: MD-OBS-A-001
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Vascular Disease, Peripheral; Chronic Wound of the Lower Limb (Leg Ulcer or Foot Ulcer)
Keywords: multispectral near-infrared spectroscopy; chronic wound; peripheral vascular disease; near-infrared imaging; ABI; tissue oxygenation; tissue oximetry; TBI; TCOM; TcPO2; Doppler
MeSH Terms: conditions — Peripheral Vascular Diseases; Leg Ulcer; Foot Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn if the measures of tissue oxygenation from the MIMOSA Pro imaging device correlate to standard vascular assessment tools in patients who receiving a lower extremity vascular assessment.

The main questions it aims to answer are:

* Do the MIMOSA Pro tissue oxygenation measures correlate to Ankle-Brachial Index, Toe-Brachial Index, transcutaneous oximetry, and Doppler wave forms?
* Do the MIMOSA Pro tissue oxygenation measures correlate with disease classifications for peripheral arterial disease, venous disease, and wound stage?
* Is the MIMOSA Pro able to measure vascular status more often than other modalities?

Participants will be asked to follow standard of care, and also allow for their legs to imaged by the MIMOSA Pro.

DETAILED DESCRIPTION:
Observational non-interventional study to assess the use of multispectral near-infrared (MS-NIR) imaging as an adjunct tool in the wound center. No clinical decisions will be made based on information obtained through the use of the MIMOSA device. Objectives are to correlate tissue oxygen saturation (StO2) by MS-NIR to measures by standard vascular diagnostic tools, including ankle-brachial index (ABI), toe-brachial index (TBI), transcutaneous oximetry, Doppler waveforms. Also to assess the ability of MS-NIR to support the classification and grading severity of patients' peripheral artery disease (PAD), venous disease and wound healing and to evaluate the clinical workflow utility of MS-NIR as an adjunct tool in the wound center. The study will recruit patients 18 years old and older, are undergoing an ankle-brachial index exam and recently had/will have further vascular assessment, as per standard of care (inc. transcutaneous oxygen pressure, Doppler waveforms). Participants will be asked to allow for imaging of their lower extremities with the MIMOSA Pro. Investigator will assess participants on their disease and wound status. They will also perform vascular assessments mentioned above as per standard of care. Participants will be followed for 2 months as per regularly scheduled visits. The standard vascular assessment results and disease/wound status will then be correlated with the measures from the MIMOSA Pro.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 and older
* Patient is undergoing an ABI test.
* Patient recently had/will have further vascular assessment, as per standard of care (inc. transcutaneous oxygen pressure, Doppler waveforms)
* Patients who can be followed by the same investigating team for the whole period of their participation in the study.

Exclusion Criteria:

* Patients who are participating in another clinical study for ulcer management
* Patients who are unable to understand the aims of the study and not able to provide informed consent
* Receiving radiation to the extremity
* Active charcot joints

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: outpatient wound center
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient between MIMOSA measures to standard vascular assessment modalities | From baseline to the end of study at 2 months

SECONDARY OUTCOMES:
Correlation coefficient between MIMOSA measures to disease and/or wound status | From baseline to the end of study at 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health Comprehensive Wound Healing Center, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No